CLINICAL TRIAL: NCT04538365
Title: Effect on the Reduction of Bacterial Load in Surgical Antisepsis of Hands After Washing With Triclosan 0.5% Compared to Propan-1-ol 60% Used as Reference Disinfectant
Brief Title: Pre-surgical Antisepsis of Hands After Washing With Triclosan 0.5% Compared to Propan-1-ol 60%
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centro Ortopedico y Quirurgico del Pie (Other)
Responsible Party: Principal Investigator, Ricardo Becerro de Bengoa Vallejo, Principal Investigator, Centro Ortopedico y Quirurgico del Pie
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RICBEC1
Record Dates: First submitted 2020-08-29; First posted 2020-09-04 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-10

CONDITIONS: Antisepsis
Keywords: hand washing; presurgical antisepsis
MeSH Terms: interventions — Triclosan; Solutions; Propranolol

STUDY DESIGN:
Intervention Model Description: Crossover design is used
Who Masked: Outcomes Assessor
Masking Description: The samples will be sent to the laboratory with numbers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hand antisepsis with propanolol-1 60% (Active Comparator): Effectiveness of pre-surgical hand washing in reducing bacterial load using propanolol-1 60% as control
  Interventions: Drug: propanolol
- Hand antisepsis with triclosan solution (Experimental): Effectiveness of pre-surgical hand washing in reducing bacterial load using triclosan 0.5% solution
  Interventions: Drug: Triclosan 0.5 % Topical Solution

INTERVENTIONS:
Drug: Triclosan 0.5 % Topical Solution — Hand antisepsis by scrub Surgical Hand scrubbing using triclosan 0.5% solution both hands using a sterile disposable surgical scrub brush with plastic bristles on one side and a foam sponge on the other side
  Other Names: Hand antisepsis with Triclosan 0.5% solution.
  Arms: Hand antisepsis with triclosan solution
Drug: propanolol — Hand antisepsis by scrub Surgical Hand scrubbing using Propanolol 60% solution both hands using a sterile disposable surgical scrub brush with plastic bristles on one side and a foam sponge on the other side
  Other Names: Hand antisepsis with Propanolol 60% solution
  Arms: Hand antisepsis with propanolol-1 60%

SUMMARY:
The present study evaluates the effects of bactericidal load reduction after surgical hand scrub antisepsis using the reference antiseptic product propanol-

1 60% as control versus a surgical hand scrub antisepsis with triclosan 0.5% in order to test if pass the standard european norm 12791.

DETAILED DESCRIPTION:
The investigators conducted a crossover clinical trial to evaluate the antiseptic effectiveness of preoperative surgical scrubbing using propan-ol-1 60% by scrub using the reference antiseptic product propan-ol-1 60% as control versus a surgical hand scrub antisepsis with trocilosan 0.5% in order to test if pass the standard european norm 12791. Samples will be taken from the hands of each volunteer after a surgical hands antiseptic.

ELIGIBILITY:
Inclusion Criteria:

* Participants without systemic pathologies, with healthy skin of the hands and short fingernails.
* They do not use substances with antibacterial action.

Exclusion Criteria:

* Taken antibiotics before 10 days of the intervention.
* Wear any jewellery on the hands

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Reduction of bacterial load immediately after hand scrub | Change from bacterial load at 5 minutes
  Participants will scrub with the antiseptic solution vigorously from hand to the wrists according with the standard handscrub procedure

SECONDARY OUTCOMES:
Reduction of bacterial load after 3 hours of hand scrub | Change from bacterial load after 3 hours
  Participants will scrub with the antiseptic solution vigorously from hand to the wrists according with the standard handscrub after 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo B Becerro de Bengoa Vallejo, PhD, Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- Facultad de Enfermeria, Fisioterapia y Podologia, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
A number will be assigned to each participant

REFERENCES:
- [Derived] Sante L, Gomez-Lus ML, Martin-Villa C, Becerro-de-Bengoa-Vallejo R, Alou L, Sevillano D. Effect on the reduction of bacterial load after surgical hand antisepsis with triclosan 0.5% compared to triclosan 0.5% followed by 70% alcoholic solution. Infect Control Hosp Epidemiol. 2023 Mar;44(3):517-519. doi: 10.1017/ice.2021.506. Epub 2021 Dec 22. PMID 34933701